CLINICAL TRIAL: NCT00010270
Title: A Phase I Study Of LMB-9, A Recombinant Disulfide Stabilized Anti-Lewis Y Immonutoxin Administered By 5-Days Continuous Infusion For Patients With Colorectal Adenocarcinoma
Brief Title: LMB-9 Immunotoxin in Treating Patients With Advanced Pancreatic, Esophageal, Stomach, Colon, or Rectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068462; UFMC-431; UFMC-IND-7697; UFMC-NSC-691236; NCI-431; EU-20120
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-01

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; stage III pancreatic cancer; stage II pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV gastric cancer; adenocarcinoma of the stomach; recurrent gastric cancer; adenocarcinoma of the esophagus; stage IV esophageal cancer; stage III esophageal cancer; recurrent esophageal cancer; stage II esophageal cancer; adenocarcinoma of the rectum; stage III colon cancer; stage III rectal cancer; stage III gastric cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Biological: LMB-9 immunotoxin

SUMMARY:
RATIONALE: LMB-9 immunotoxin can locate tumor cells and kill them without harming normal cells. This may be an effective treatment for advanced pancreatic, esophageal, stomach, colon or rectal cancer.

PURPOSE: Phase I trial to study the effectiveness of LMB-9 immunotoxin in treating patients who have advanced pancreatic, esophageal, stomach, colon, or rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of LMB-9 immunotoxin in patients with advanced adenocarcinoma of the colon, rectum, pancreas, esophagus, or stomach with overexpression of the Lewis-Y antigen.
* Determine the maximum tolerated dose of this drug in these patients.
* Determine the clinical response of patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive LMB-9 immunotoxin IV continuously on days 1-5. Patients with stable or responding disease after completion of the first course receive additional courses every 4-5 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of LMB-9 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 40-50 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced adenocarcinoma of the colon, rectum, pancreas, esophagus, or stomach that is refractory to standard treatment
* Overexpression of the Lewis-Y antigen
* Measurable or evaluable disease
* No CNS metastasis
* Metastatic liver disease from primary tumor allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* Absolute granulocyte count greater than 1,200/mm^3

Hepatic:

* Bilirubin normal
* SGOT and SGPT no greater than 1.5 times upper limit of normal
* Hepatitis B or C antigen negative
* No liver disease (e.g., alcohol liver disease)
* Albumin at least 3.0 g/dL

Renal:

* Creatinine no greater than 1.4 mg/dL
* Creatinine clearance at least 60 mL/min
* Proteinuria no greater than 1 g/24 hours (grade II toxicity-like)

Cardiovascular:

* No prior coronary artery disease
* No New York Heart Association class II, III, or IV congestive heart failure
* No arrhythmia requiring treatment

Pulmonary:

* FEV_1 and FVC greater than 65% predicted

Other:

* No other concurrent malignancy
* No active peptic ulcer disease
* No known allergy to omeprazole
* No known seizure disorder
* No concurrent medical or psychiatric condition that would preclude study participation
* No contraindication to pressor therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hafkemeyer, MD, Study Chair — Kreiskrankenhaus Emmendingen
Locations (1):
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany